CLINICAL TRIAL: NCT06178380
Title: Clinical and Instrumental Biomechanical Assessement and Rehabilitation of Patients With Knee Osteoarthritis:A Randomized Single Blind Clinical Trial
Brief Title: Instrumental Versus Standard Rehabilitation for Knee Osteoarthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mohammed V Souissi University (Other)
Collaborators: Ibn Sina University Hospital, Rabat, Morocco (Other)
Responsible Party: Principal Investigator, EL Moudane Houda, principal Investigator, Mohammed V Souissi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: knee osteoarthritis
Record Dates: First submitted 2023-11-03; First posted 2023-12-21 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2023-12

CONDITIONS: Knee Osteoarthritis
Keywords: rehabilitation; knee; osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — Rehabilitation

STUDY DESIGN:
Intervention Model Description: A randomized single blind clinical trial is a research study design used to evaluate the effectiveness of a medical intervention or treatment. In this type of trial, participants are randomly assigned to one of two a more groups, one groupe receives the experimental treatment, while the other group may receive a placebo or standard treatment, depending on the study's design
  - the term "single blind" refers to the fact that , in this trial the participants do not know whether they are receiving the experimental treatment or a control treatment this is done to minimize the potential for bias in reporting their symptoms or outcomes
Who Masked: Participant
Masking Description: Masking is a technique used to keep treatment information indisclosed to the study participants while allowing researchers and treatment administration to know this information: study participants are not informed about the treatment they are receiving, they do not know whether they are receiving the experimental treatment under investigation or if they are in the control group , which may receive a placebo or standard treatment .
  This helps reduce potential bias related to participant expectations
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard rehabilitation (Active Comparator): rehabilitation of knee osteoarthritis patients using standard techniques of massage, stretching, muscle strengthening and balance work
  Interventions: Other: rehabilitation
- instrumental rehabilitation (Experimental): rehabilitation of knee osteoarthritis patients using isokinetic, posturograph and antigravity treadmill
  Interventions: Other: rehabilitation

INTERVENTIONS:
Other: rehabilitation — For the experimental group:
  Isokinetic training Antigravity treadmill Posturography
  For the control group:
  Patients will receive a standard rehabilitation prescription comprising:
  Physiotherapy , muscle stretching and strengthening , proprioceptive exercises, and self-programmed

SUMMARY:
A randomized clinical trial to evaluate the effectiveness of an instrumental rehabilitation protocol compared with standard protocol In patients with knee osteoarthritis.

DETAILED DESCRIPTION:
This is a randomized clinical trial designed to compare two intervention aimed at reducing and improving knee function in patients with knee osteoarthritis

- sixty subjects suffering from knee osteoarthritis will be recruited; 30 per group.

A: instrumental rehabilitation B:standard rehabilitation All patients who meet the clinical inclusion and exclusion criteria will have a standard radiography

* selected patients will be invited to participate and will be informed of the purpose and conduct of the study
* patients will be randomized to either the instrumental rehabilitation programme groupe or the standard rehabilitation group
* patients in both groups will have a protocol that will be extended over 6 weeks
* participants will be assessed primarily for function and pain, as well as other secondary endpoints , at baseline at 3 weeks and at 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* patients with radiologically confirmed uni/ bilateral gonarthrosis

Exclusion Criteria:

* Will be excluded from our study:
* Subjects with congestive gonarthrosis (joint effusion at clinical examination).
* Patients followed for chronic inflammatory rheumatism.
* Patients who are candidates for surgery for knee osteoarthritis
* Patients with a pathology causing a limitation in walking distance apart from gonarthrosis.
* Amputees of one or both lower limbs.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Le Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | 12 weeks
  The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) is an assessment tool developed to measure pain, stiffness, and physical function in individuals with osteoarthritis, primarily in the knee and hip. Patients' responses to each question are typically scored on a scale ranging from 0 to 4, where 0 signifies "no symptoms" and 4 signifies "severe symptoms." Scores obtained in each subscale can be combined to provide a total score or used individually to assess specific aspects of osteoarthritic symptoms.

SECONDARY OUTCOMES:
Joint amplitude measurements | 12 weeks
  using a goniometer to evaluate the extent of knee flexion and extension
muscle testing of hamstring and quadriceps | 12 weeks
  Muscle testing is employed to assess hamstring and quadriceps strength on a qualitative scale ranging from 0 to 5
time up and go | 12 weeks
  is utilized to evaluate patient mobility and balance, measured in seconds,Less than 13.5 seconds: Low risk of falling; the person has good walking speed and functional mobility.
  13.5 seconds or more: High risk of falling; the person does not have good walking speed or functional mobility.
the Visual Analog Scale | 12 weeks
  the Visual Analog Scale (VAS), a graded scale ranging from 0 to 100 millimeters, 0 no pain and 100 severe pain
quality of life index | 12 weeks
  the SF12 questionnaire is administered to assess quality of life,The minimum value is 0, and the maximum value is 100,Scores above 50 indicate a better-than-average health-related quality of life, while scores below 50 suggest below-average health.
results of balance plateform assessement | 12 weeks
  the surface area of the confidence ellipse in square millimeters , length of the stabilogram in millimeters, x and y coordinates of the center of pressure in millimeters
muscle testing of hamstring and quadriceps using an isokinetic dynamometer | 12 weeks
  peak torque in newtons and body weight in newtons per kilogram
walking test | 12 weeks
  support symmetry in percentage and step length in centimeters

CONTACTS AND LOCATIONS:
Overall Officials: Houda EL Moudane, phd student, Principal Investigator — Mohammed V Souissi University; Samia KARKOURI, PROFESSOR, Study Director — Mohammed V Souissi University; Latifa TAHIRI, PROFESSOR, Study Director — Mohammed V Souissi University; Sara SKALLI, Doctor, Study Chair — Mohammed V Souissi University
Locations (2):
- Morocco (2):
  - Houda EL Moudane, Rabat
  - Houda EL Moudane, Salé

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lespasio MJ, Piuzzi NS, Husni ME, Muschler GF, Guarino A, Mont MA. Knee Osteoarthritis: A Primer. Perm J. 2017;21:16-183. doi: 10.7812/TPP/16-183. PMID 29035179
- See also: on this site we will find the definition of osteoarthritis of the knee and the risk factors as well as the diagnosis and treatment of this pathology — https://www.passeportsante.net/fr/Maux/Problemes/Fiche.aspx?doc=gonarthrose